CLINICAL TRIAL: NCT05910840
Title: Support-t, an Online Training and Peer Support Platform to Accompany Youth Living With Type 1 Diabetes Transitioning to Adult Healthcare
Brief Title: Support-t Online Training in Youth Living With Type 1 Diabetes Transitioning to Adult Care
Acronym: Support-t
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anne-Sophie Brazeau (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other); CSSS de Gatineau (Other); Centre de recherche du CHU de Sherbrooke (Unknown); CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor-Investigator, Anne-Sophie Brazeau, Associate Professor, McGill University
Organization: McGill University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MP-37-2024-9734
Record Dates: First submitted 2023-06-06; First posted 2023-06-20 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders (Including Diabetes Mellitus); Metabolic Disease; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases
Keywords: Transition Care; Pediatric; Adolescent; Education; Hemaglobin A1c; Self-management; Randomized Controlled Trial
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases; Autoimmune Diseases; Immune System Diseases

STUDY DESIGN:
Intervention Model Description: Active arm: Participants randomized to the active arm will have access to the Support-t online training and peer support platform in addition to their usual diabetes care, over the 18 month intervention period. Support-t contains 3 components: 1) Educational material, 2) News blog and 3) Patients' discussion forum.
  Control arm: Participants randomized to usual care only will attend their usual diabetes clinic visits, over the 18-month intervention period, which consists of visits with their health care provider and ad-hoc diabetes education with nurses and dietitians.
Who Masked: Outcomes Assessor
Masking Description: Data analysts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Support-t plus usual diabetes care (Experimental): Access to the Support-t online training and peer support platform in addition to usual diabetes care for 18 months. Support-t contains 3 components: 1) Educational material, 2) News blog and 3) Patients' discussion forum. Health care providers from the pediatric diabetes clinics will receive Support-t training and will be encouraged to recommend the Support-t platform during routine care with their patients from the active arm.
  Interventions: Other: Support-t
- Usual diabetes care only (No Intervention): Usual diabetes care for 18 months, which consists of visits with their health care provider and ad-hoc diabetes education with nurses and dietitians. Health care providers from the pediatric diabetes clinics will be instructed not to discuss or refer to the Support-t platform with patients from the control arm. Control arm participants will have the option to use the Support-t platform after the 18-month study.

INTERVENTIONS:
Other: Support-t — Support-t plus usual diabetes care for 18 months
  Arms: Support-t plus usual diabetes care

SUMMARY:
The investigators will conduct a randomized controlled trial (RCT) to examine how an online training and peer support platform could help the preparation to transition to adult care. Among 14-16 year old youth with Type 1 Diabetes (T1D), the investigators aim to assess the effect of an online training and peer support platform (Support-t) integrated in usual care, compared with usual care on Hemoglobin A1c (HbA1c), adverse outcomes and psychosocial measures during the preparation for transition to adult care. The investigators will conduct a multi-site, parallel group, blinded (outcome assessors, data analysts), superiority RCT of adolescents with T1D (14-16 years of age) followed at one of 4 university teaching hospital-based pediatric diabetes clinics in the province of Quebec.

DETAILED DESCRIPTION:
The transition from pediatric to adult diabetes care is a challenging period for adolescents and young adults living with chronic conditions, such as Type 1 Diabetes (T1D). For youth with T1D, transition from pediatric to adult care is characterized by deterioration in glycemic control (Hemoglobin A1c [HbA1c]), reduced adherence to diabetes management tasks and increased risk of diabetes complications. The investigators propose to examine an online training and peer support platform as a potential alternative for delivering transition care. In adolescents with T1D, the investigators hypothesize that an online training and peer support platform (Support-t), when integrated into usual pediatric care, as compared with usual care alone, will result in better HbA1c, less adverse outcomes and better psychosocial outcomes during the preparation for transfer to adult care.

Primary Aim: To determine the impact of adding access to Support-t to usual care compared with usual care alone, on HbA1c during the preparation for transfer to adult care.

Secondary Aims: To determine the impact of adding access to Support-t to usual care compared with usual care alone, on self-efficacy, diabetes distress, quality of life (QOL; diabetes specific), readiness to transfer to adult care, glucose management, severe hypoglycemic episodes, diabetic ketoacidosis (DKA), T1D-related ED-visits and hospitalizations during the preparation for transfer to adult care. 2. To determine the cost-effectiveness of Support-t. 3. To understand the context for implementation in regards to level of engagement on Support-t, satisfaction and experience (barriers, facilitators) with Support-t.

Methods: The investigators will conduct a multi-site, parallel group, blinded (outcome assessors, data analysts), superiority RCT of adolescents with T1D (14-16 years of age) followed at one of 4 university teaching hospital-based pediatric diabetes clinics in Quebec. Patients will be recruited over 20 months. Interventions will occur over 18 months. Follow-up will be to 18 months from enrollment. Allocation will be concealed with a 1:1 intervention to control ratio. Participants in the active arm will have access to a mobile-based online training and peer support platform (Support-t) added to usual care. Participants in the control group will have in parallel with the intervention group, their usual diabetes care. The primary outcome is the change in HbA1c measured at 18 months (HbA1c measured at 18 months - HbA1c measured at baseline). Secondary outcomes are self-efficacy, diabetes distress, QOL, readiness to transfer, glucose management, severe hypoglycemic episodes, DKA, T1D-related ED-visits and hospitalizations. Assessments are at baseline, 6, 12 and 18 months. Analysis will be by intention-to-treat. Outcomes will be calculated and compared between the 2 trial arms using differences with 95% Confidence Intervals, along with a cost-effectiveness analysis. Interviews will be conducted to analyze the context for implementation.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with a clinical diagnosis of T1D
* 14-16 years of age
* Receiving diabetes care at one of 4 university teaching hospital-based pediatric diabetes clinics in Quebec: Montreal Children's Hospital-McGill University Health Centre, Centre hospitalier universitaire de Sherbrooke, Le Copain-Hôpital de Gatineau, Centre Hospitalier Universitaire de Québec
* Having access to internet
* Having an active email address
* Fluent in English or French

Exclusion Criteria:

* Severe neurocognitive disabilities
* Patients with conditions associated with shortened erythrocyte survival, such as hemolytic anemia or other conditions associated with inaccurate HbA1c

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Hemaglobin A1c (HbA1c) at 18 months | 18 months
  HbA1c measured with a venous or capillary blood sample as part of the standard of diabetes care will be derived from the medical record chart or measured using an A1c Test Kit, which is a non-fasting, finger prick, whole blood test

SECONDARY OUTCOMES:
Change from Baseline Hemaglobin A1c (HbA1c) at 6 and 12 months | 6, 12 months
  HbA1c measured with a venous or capillary blood sample as part of the standard of diabetes care will be derived from the medical record chart or measured using an A1c Test Kit, which is a non-fasting, finger prick, whole blood test
Continuous Glucose Monitoring (CGM) - % Time in range | 0, 6, 12, 18 months
  % Time in range (3.9-10.0mmol/L) over the past 4 weeks will be derived from the medical record chart
Continuous Glucose Monitoring (CGM) - % Time above range | 0, 6, 12, 18 months
  % Time above range (3.9-10.0mmol/L) over the past 4 weeks will be derived from the medical record chart
Continuous Glucose Monitoring (CGM) - % Time below range | 0, 6, 12, 18 months
  % Time below range (3.9-10.0mmol/L) over the past 4 weeks will be derived from the medical record chart
Continuous Glucose Monitoring (CGM) - Standard deviation | 0, 6, 12, 18 months
  Standard deviation of the past 4 weeks will be derived from the medical record chart
Continuous Glucose Monitoring (CGM) - % Coefficient of variation | 0, 6, 12, 18 months
  % Coefficient of variation of the past 4 weeks will be derived from the medical record chart
Severe hypoglycemic events | 0, 6, 12, 18 months
  Any severe hypoglycemic events in the past 6 months will be derived from self-report and from the medical record chart
Diabetic Ketoacidosis (DKA) events | 0, 6, 12, 18 months
  Any Diabetic Ketoacidosis (DKA) events in the past 6 months will be derived from self-report and from the medical record chart
Diabetes-related hospitalizations | 0, 6, 12, 18 months
  Any diabetes-related hospitalizations in the past 6 months, expressed as number of hospitalizations per person-years (P-Y) at risk will be derived from self-report and from the medical record chart
Diabetes-related emergency department visits | 0, 6, 12, 18 months
  Any diabetes-related emergency-department visits in the past 6 months, expressed as number of emergency department visits per person-years (P-Y) at risk will be derived from self-report and from the medical record chart
Self-efficacy | 0, 6, 12, 18 months
  Self-efficacy for Diabetes Self-Management Measure (SEDM) assesses self-efficacy. The score ranges from 1 to 10. All item scores are averaged to compute the score. A higher score represents a better outcome.
Diabetes distress | 0, 6, 12, 18 months
  Problem Areas in Diabetes Scale-Teen (PAID-T) assesses adolescent diabetes distress. The scores range from 14 to 84. A total distress score is computed by summing responses. Higher scores indicate youth perception of feeling more burdened related to T1D.
Diabetes specific Quality of Life (QOL) | 0, 6, 12, 18 months
  Type 1 Diabetes and Life (T1DAL) questionnaire assesses diabetes specific QOL for 12-17 year old adolescents living with T1D. Scores are transformed on a scale from 0 to 100. The total score ranges from 0 to 100. To calculate the total score, the mean is computed as the sum of all item scores divided by the number of items answered on all the scales. A higher total score represents a better outcome. The subscale scores (Daily Emotional Experiences & Daily Activities, Handling Diabetes Well, Peer Relationships, and Family Relationships) range from 0 to 100. To calculate the subscale scores, the mean is computed as the sum of the items in the subscale divided by the number of items answered on the subscale. Higher subscale scores represent a better outcome.
Transition readiness | 0, 6, 12, 18 months
  Readiness Assessment of Emerging Adults with Type 1 Diabetes Diagnosed in Youth (READDY) assesses diabetes-related knowledge or skill items by querying respondents on 42 total items split into 5 domains: knowledge, navigation, health behaviors, and insulin pump skills. Respondents answer on a Likert scale from "yes, I can do this" scored 5 to "Haven't thought about it" scored 1. Confidence level is evaluated in each domain with a higher score indicating more confidence.
Cost effectiveness (HbA1c) | 12 and 18 months
  Cost effectiveness of access to Support-t in addition to usual care compared with usual care in terms of incremental cost effectiveness ratio (ICER) for HbA1c
Cost effectiveness (self-efficacy) | 12 and 18 months
  Cost effectiveness of access to Support-t in addition to usual care compared with usual care in terms of incremental cost effectiveness ratio (ICER) for self-efficacy
Cost effectiveness (diabetes distress) | 12 and 18 months
  Cost effectiveness of access to Support-t in addition to usual care compared with usual care in terms of incremental cost effectiveness ratio (ICER) for diabetes distress
Cost effectiveness (QOL) | 12 and 18 months
  Cost effectiveness of access to Support-t in addition to usual care compared with usual care in terms of incremental cost effectiveness ratio (ICER) for QOL

OTHER OUTCOMES:
Engagement with Support-t platform (T1D patient) - time in minutes on platform | 6, 12, 18 months
  Engagement metrics will be extracted using Google analytics - time (minutes) spent on the platform
Engagement with Support-t platform (T1D patient) - discussion forum participation | 6, 12, 18 months
  Engagement metrics will be extracted using Google analytics - participation on the platform discussion forum
Engagement with Support-t platform (T1D patient) - content accessed | 6, 12, 18 months
  Engagement metrics will be extracted using Google analytics - specific content accessed from the platform
Engagement with Support-t platform (T1D patient) - total pages viewed | 6, 12, 18 months
  Engagement metrics will be extracted using Google analytics - total pages viewed from the platform
Engagement with Support-t platform (T1D patient) - downloaded documents | 6, 12, 18 months
  Engagement metrics will be extracted using Google analytics - downloaded documents from the platform
Engagement with Support-t platform (T1D patient) - use of calculators | 6, 12, 18 months
  Engagement metrics will be extracted using Google analytics - use of calculators on the platform
Engagement with Support-t platform (Health Care Provider) - time in minutes on platform | 6, 12 months
  Engagement metrics will be extracted using Google analytics - time (minutes) spent on the platform
Engagement with Support-t platform (Health Care Provider) - content accessed | 6, 12 months
  Engagement metrics will be extracted using Google analytics - specific content accessed from the platform
Engagement with Support-t platform (Health Care Provider) - total pages viewed | 6, 12 months
  Engagement metrics will be extracted using Google analytics - total pages viewed from the platform
Engagement with Support-t platform (Health Care Provider) - downloaded documents | 6, 12 months
  Engagement metrics will be extracted using Google analytics - downloaded documents from the platform
Engagement with Support-t platform (Health Care Provider) - use of calculators | 6, 12 months
  Engagement metrics will be extracted using Google analytics - use of calculators on the platform
Satisfaction with Support-t platform - T1D patient | 6, 12, 18 months
  Satisfaction will be rated on a scale from 1 to 10. Higher scores indicate greater satisfaction with the platform.
Experience with Support-t platform (Barriers, facilitators, satisfaction, fidelity) - T1D patient | 18 months
  Individual interviews to understand the experience in the context of implementation of the Support-t platform (Barriers, facilitators, satisfaction, fidelity) using qualitative descriptive methodology
Experience with Support-t platform (Barriers, facilitators, satisfaction, fidelity) - Health Care Provider | 12 months
  Individual interviews to understand the experience in the context of implementation of the Support-t platform (Barriers, facilitators, satisfaction, fidelity) using qualitative descriptive methodology

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Brazeau, PhD, Principal Investigator — School of Human Nutrition - McGill University
Locations (4):
- Canada (4):
  - Clinique de pédiatrie Le Copain-Hôpital de Gatineau, Gatineau
  - Montreal Children's Hospital - McGill University Health Centre, Montreal
  - Centre Hospitalier Universitaire de Québec, Québec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke

REFERENCES:
- [Background] Sanmugalingham G, Mok E, Cafazzo JA, Desveaux L, Brazeau AS, Booth GL, Greenberg M, Kichler J, Rac VE, Austin P, Goldbloom E, Henderson M, Landry A, Zenlea I, Taylor M, Nakhla M, Shulman R. Text message-based intervention, Keeping in Touch (KiT), to support youth as they transition to adult type 1 diabetes care: a protocol for a multisite randomised controlled superiority trial. BMJ Open. 2023 May 8;13(5):e071396. doi: 10.1136/bmjopen-2022-071396. PMID 37156577
- [Background] Xie LF, Housni A, Nakhla M, Cianci R, Leroux C, Da Costa D, Brazeau AS. Adaptation of an Adult Web Application for Type 1 Diabetes Self-management to Youth Using the Behavior Change Wheel to Tailor the Needs of Health Care Transition: Qualitative Interview Study. JMIR Diabetes. 2023 Apr 26;8:e42564. doi: 10.2196/42564. PMID 37121571
- [Background] Ladd JM, Reeves-Latour J, Dasgupta K, Bell LE, Anjachak N, Nakhla M. Toward a better understanding of transition from paediatric to adult care in type 1 diabetes: A qualitative study of adolescents. Diabet Med. 2022 May;39(5):e14781. doi: 10.1111/dme.14781. Epub 2022 Jan 7. PMID 34967058
- [Background] Mok E, Henderson M, Dasgupta K, Rahme E, Hajizadeh M, Bell L, Prevost M, Frei J, Nakhla M. Group education for adolescents with type 1 diabetes during transition from paediatric to adult care: study protocol for a multisite, randomised controlled, superiority trial (GET-IT-T1D). BMJ Open. 2019 Nov 11;9(11):e033806. doi: 10.1136/bmjopen-2019-033806. PMID 31719096
- [Background] Alwadiy F, Mok E, Dasgupta K, Rahme E, Frei J, Nakhla M. Association of Self-Efficacy, Transition Readiness and Diabetes Distress With Glycemic Control in Adolescents With Type 1 Diabetes Preparing to Transition to Adult Care. Can J Diabetes. 2021 Jul;45(5):490-495. doi: 10.1016/j.jcjd.2021.05.006. Epub 2021 May 19. PMID 34176613
- [Background] Michaud S, Dasgupta K, Bell L, Yale JF, Anjachak N, Wafa S, Nakhla M. Adult care providers' perspectives on the transition to adult care for emerging adults with Type 1 diabetes: a cross-sectional survey. Diabet Med. 2018 Jul;35(7):846-854. doi: 10.1111/dme.13627. Epub 2018 May 2. PMID 29577410
- [Background] Lafontaine S, Mok E, Frei J, Henderson M, Rahme E, Dasgupta K, Nakhla M. Associations of Diabetes-related and Health-related Quality of Life With Glycemic Levels in Adolescents With Type 1 Diabetes Preparing to Transition to Adult Care. Can J Diabetes. 2023 Aug;47(6):525-531. doi: 10.1016/j.jcjd.2023.05.002. Epub 2023 May 12. PMID 37182591
- [Background] Soufi A, Mok E, Henderson M, Dasgupta K, Rahme E, Nakhla M. Association of stigma, diabetes distress and self-efficacy with quality of life in adolescents with type 1 diabetes preparing to transition to adult care. Diabet Med. 2024 Jan;41(1):e15159. doi: 10.1111/dme.15159. Epub 2023 Jun 21. PMID 37269172
- [Background] Wafa S, Nakhla M. Improving the Transition from Pediatric to Adult Diabetes Healthcare: A Literature Review. Can J Diabetes. 2015 Dec;39(6):520-8. doi: 10.1016/j.jcjd.2015.08.003. Epub 2015 Oct 20. PMID 26498219
- [Background] Nakhla M, Daneman D, To T, Paradis G, Guttmann A. Transition to adult care for youths with diabetes mellitus: findings from a Universal Health Care System. Pediatrics. 2009 Dec;124(6):e1134-41. doi: 10.1542/peds.2009-0041. Epub 2009 Nov 23. PMID 19933731
- [Background] Nakhla M, Daneman D, Frank M, Guttmann A. Translating transition: a critical review of the diabetes literature. J Pediatr Endocrinol Metab. 2008 Jun;21(6):507-16. PMID 18717235
- [Background] Nakhla M, Bell LE, Wafa S, Dasgupta K. Improving the transition from pediatric to adult diabetes care: the pediatric care provider's perspective in Quebec, Canada. BMJ Open Diabetes Res Care. 2017 Jun 30;5(1):e000390. doi: 10.1136/bmjdrc-2017-000390. eCollection 2017. PMID 28761657
- [Background] Robinson ME, Simard M, Larocque I, Shah J, Rahme E, Nakhla M. Psychiatric disorders in emerging adults with diabetes transitioning to adult care: A retrospective cohort study. Diabet Med. 2021 Jun;38(6):e14541. doi: 10.1111/dme.14541. Epub 2021 Feb 19. PMID 33576092
- [Derived] Roy-Fleming A, Nakhla M, Mok E, Vanasse A, Cianci L, Kichler J, Simoneau-Roy J, Couture Y, Gagne J, Dupont M, Brazeau AS. Support-t, an online training and peer support platform to accompany youth living with type 1 diabetes transitioning to adult healthcare: protocol of an effectiveness-implementation trial. BMJ Open. 2025 Oct 6;15(10):e105514. doi: 10.1136/bmjopen-2025-105514. PMID 41057177